CLINICAL TRIAL: NCT00526058
Title: Randomized Multicenter Crossover Study to Compare the Plasmat® Futura Heparin Induced Extracorporeal Lower Density Lipo-Protein (LDL) Precipitation (H.E.L.P.) Apheresis System to the Approved Secura System in the Reduction of LDL-c in Patients With Hypercholesterolemia
Brief Title: (H.E.L.P.)Apheresis Therapy to Compare the Reduction of LDL (Low Density Lipoprotein) Cholesterol
Acronym: FUTURA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LDLc-A-US2-0406
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Results first posted 2010-07-30 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Hypercholesterolemia
Keywords: Heparin; Extracorporeal; Low Density Lipo-Protein (LDL) Cholesterol; Apheresis; Device
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Secura then Futura) (Other): The Group Randomized first to the approved Plasmat® Secura apheresis system and then to the Plasmat® Futura apheresis system.
  Interventions: Device: Secura then Futura
- B (Futura then Secura) (Other): The Group Randomized first to the approved Plasmat® Futura apheresis system and then to the Plasmat® Secura apheresis system.
  Interventions: Device: Futura then Secura

INTERVENTIONS:
Device: Secura then Futura — Randomized to 6 bi-monthly H.E.L.P. therapy treatments with the Plasmat® Secura apheresis system and then cross over to receive 6 bi-monthly treatments with the Plasmat® Futura apheresis system.
  Arms: A (Secura then Futura)
Device: Futura then Secura — Randomized to 6 bi-monthly H.E L.P. therapy treatments with the Plasmat® Futura apheresis system and then cross over to receive 6 bi-monthly treatments with the Plasmat® Secura apheresis system.
  Arms: B (Futura then Secura)

SUMMARY:
The primary objective of the study is to demonstrate that the performance of the modified Plasmat® Futura H.E.L.P. Apheresis System is non-inferior to the current FDA approved Plasmat® Secura H.E.L.P Apheresis System for use under the approved indication of the acute reduction of LDL-cholesterol from the plasma in populations for whom diet has been ineffective and maximum drug therapy has either been ineffective or not tolerated.

DETAILED DESCRIPTION:
The primary study endpoint is the change in percent measurements of the pre-to-post apheresis LDL measurements between the approved H.E.L.P. system and the modified H.E.L.P. system. The secondary study endpoints are clinical lab profiles and device parameters analyzed at specific time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 25 and 70 years of age (inclusive) at the time of randomization.
* Subject is an appropriate candidate for H.E.L.P. apheresis treatment for hypercholesterolemia according to current Plasmat® Secura approval criteria.
* Subject has received a minimum of two consecutive bi-monthly* H.E.L.P. apheresis treatments using the Plasmat® Secura apheresis system >30 days prior to the screening visit.
* Subject is willing to maintain cholesterol lowering dietary and drug therapies as prescribed through the course of the study.
* Subject is willing and able to provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) Waiver.
* Sterile, post-menopausal, or using acceptable birth control for the duration of the study. Acceptable birth control is defined as having a vasectomized, postmenopausal, or sterile partner; the ongoing use of approved hormonal contraceptives, barrier method, or an intrauterine device; or abstinence.

  * Every 14 days (±2 days)

Exclusion Criteria:

* A History of a known sensitivity to heparin or ethylene oxide.
* A history of hemorrhagic diathesis, bleeding/clotting disorder, thrombocytopenia (defined as platelet count < 150 x109/L), or for whom the use of heparin would cause excessive or uncontrolled anticoagulation or for whom adequate anticoagulation cannot be safely achieved (ie., hemophilia, recent surgery, acute internal bleeding, gastrointestinal ulcers).
* Females who are pregnant or lactating.
* Subjects< 106 lbs. or <48.2 kg in body weight; or whose weight is >1.5 times their ideal weight.
* Certain cardiac impairments such as congestive heart failure, major arrhythmia, or diastolic blood pressure greater than 100 mm/Hg on two separate occasions at least 24 hours apart.
* Renal insufficiency defined as creatinine greater >2.0 mg/dlL or is dependent upon renal dialysis.
* Untreated hypothyroidism; uncontrolled diabetes mellitus; or fasting triglycerides >500 mg/dL.
* Serious systemic disease (e.g., advanced neoplasms, and acute hepatitis) including Immune system suppression or compromise, that could preclude survival to study completion.
* History of stroke within 6 months of the screening visit.
* Received thrombolytic treatment < 7 days of screening.visit.
* Taken or requires a prohibited treatment < 30 days prior to the Screening Visit, or requires a prohibited treatment at anytime during the course of the study.
* Neutropenia (neutrophil count < 0.5 x109/L).
* History of liver disease or serum ALT and/or AST > 2X upper limit of normal range.
* History of dementia.
* History of anemia (value outside the lower normal range).
* acetyl salicylic acid (ASA) > 325 mg/day.
* Subject currently enrolled in another investigational study (does not apply to PMS for Secura device).
* Subject with any other medical condition that in the opinion of the investigator might put the subject at risk or interfere with his/her participation.
* Subject is unwilling or unable to comply with the protocol or to cooperate fully with the investigator or site personnel.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Moriarty, M.D., Principal Investigator — University of Kansas Medical Center; Paul Thompson, M.D., Principal Investigator — Hartford Hospital
Locations (2):
- United States (2):
  - Hartford Hospital, Hartford, Connecticut
  - University of Kansas Medical Center, Kansas City, Kansas

REFERENCES:
- [Background] Julius U, Metzler W, Pietzsch J, Fassbender T, Klingel R. Intraindividual comparison of two extracorporeal LDL apheresis methods: lipidfiltration and HELP. Int J Artif Organs. 2002 Dec;25(12):1180-8. doi: 10.1177/039139880202501210. PMID 12518963
- [Background] Susca M. Heparin-Induced extracorporeal low-density lipoprotein precipitation futura, a new modification of HELP apheresis: technique and first clinical results. Ther Apher. 2001 Oct;5(5):387-93. doi: 10.1046/j.1526-0968.2001.00371.x. PMID 11778925
- [Background] Schettler V, Monazahian M, Wieland E, Thomssen R, Muller GA. Effect of heparin-induced extracorporeal low-density lipoprotein precipitation (HELP) apheresis on hepatitis C plasma virus load. Ther Apher. 2001 Oct;5(5):384-6. doi: 10.1046/j.1526-0968.2001.00374.x. PMID 11778924
- [Background] Moriarty PM, Gibson CA, Shih J, Matias MS. C-reactive protein and other markers of inflammation among patients undergoing HELP LDL apheresis. Atherosclerosis. 2001 Oct;158(2):495-8. doi: 10.1016/s0021-9150(01)00633-5. PMID 11583732

RESULTS

PARTICIPANT FLOW:
Groups:
- Secura: Randomized first to the approved Plasmat® Secura apheresis system then Plasmat® Futura apheresis system.
- Futura: Randomized first to the approved Plasmat® Futura apheresis system then Plasmat® Secura apheresis system.
Period: Period: First Intervention
Arm/Group | Secura | Futura
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Period: Second Intervention
Arm/Group | Secura | Futura
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secura | Futura | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (7.76) | 59.7 (9.15) | 58.3 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Pre- and Post-treatment Reductions of Low-density Lipoprotein Cholesterol (LDL-C) Levels Between the Approved H.E.L.P. System and the Modified H.E.L.P. System.
Time Frame: Blood samples for LDL-cholesterol determination will be obtained before and after each treatment from week 0 to week 24..
Measure: Mean (90% Confidence Interval); unit: percent change
Groups:
- Secura; Futura: Data for all 18 subjects; regardless of treatment sequence (Secura-Futura or Futura-Secura)
Arm/Group | Secura | Futura
Number analyzed (Participants) | 18 | 18
percent change | 55.28 [38.6 to 71.9] | 52.89 [33.3 to 64.0]

2. Primary Outcome: Percent Change of the Pre and Post Treatment Value
Description: The primary study endpoint is the change in percent measurements of the pre-to-post apheresis LDL measurements. Blood samples for LDL-cholesterol determination will be obtained before and after each treatment. The pooled difference between the pre- and post-treatment LDL level for each apheresis machine will be reported as the primary endpoint for the system performance.
Time Frame: Assessment based on LDL-C values obtained pre-and post-treatment, analyzed from week 0 to week 24.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Secura | Futura
Number analyzed (Participants) | 18 | 18
percent change | 55.28 (9.783) | 52.89 (8.228)
Statistical Analysis 1: Comparison: Secura vs Futura; Test type: Non-Inferiority or Equivalence — Noninferiority of the Futura system to the Secura system would be demonstrated if the upper bound of the 90% confidence interval (CI) for the difference between the two systems (Secura-Futura) in percent change of LDL-C measurements from pre- to post-treatment is less than the noninferiority margin 5.7%; p = 0.005, ANOVA

3. Secondary Outcome: Clinical Lab Profiles (Pre- and Post-Treatment)
Description: Changes in pre- and post-treatment levels of total cholesterol, high-density lipoprotein cholesterol (HDL-C), total triglycerides, lipoprotein (a), fibrinogen, and C-reactive protein.
Time Frame: Analyzed at specific time points throughout the study from week 0 to week 24.
Population: Data for all 18 subjects; regardless of treatment sequence
Measure: Mean (90% Confidence Interval); unit: percent change
Arm/Group | Secura | Futura
Number analyzed (Participants) | 18 | 18
percent change
  Total Triglycerides | 63.17 [40.1 to 77.1] | 71.46 [40.8 to 89.4]
  Total Cholesterol | 50.23 [40.4 to 62.0] | 48.12 [34.6 to 59.4]
  HDL-C | 11.82 [5.6 to 19.2] | 7.41 [-3.8 to 15.4]
  VLDL-C | 62.14 [16.5 to 76.3] | 62.65 [-13.2 to 89.2]
  Lipoprotein (a) | 59.25 [43.5 to 74.4] | 49.68 [-19.5 to 74.1]
  Fibrinogen | 54.81 [38.0 to 70.8] | 52.00 [30.9 to 61.4]
  C-Reactive Protein | 58.59 [45.2 to 67.7] | 48.88 [35.0 to 59.5]

4. Secondary Outcome: Device Parameters
Description: Comparison of plasma flow rate recorded with both systems before treatment, after 500 mL of plasma treated, and at the end of each treatment session.
Time Frame: Analyzed at specific time points throughout the study from week 0 to week 24.
Population: Data for all 18 subjects; regardless of treatment sequence
Measure: Mean (Standard Deviation); unit: flow rate (mL/min)
Arm/Group | Secura | Futura
Number analyzed (Participants) | 18 | 18
flow rate (mL/min)
  Start of Session; Session 1 | 27.11 (9.380) | 12.39 (5.203)
  Start of Session; Session 2 | 23.41 (10.978) | 8.89 (4.310)
  Start of Session; Session 3 | 28.00 (13.711) | 9.67 (3.664)
  Start of Session; Session 4 | 26.35 (8.838) | 9.17 (5.079)
  Start of Session; Session 5 | 26.29 (6.049) | 10.12 (3.998)
  Start of Session; Session 6 | 27.61 (7.920) | 8.39 (3.898)
  After 500mL; Session 1 | 33.67 (6.380) | 23.44 (2.895)
  After 500mL; Session 2 | 32.59 (5.938) | 22.50 (3.552)
  After 500mL; Session 3 | 31.61 (4.354) | 22.71 (3.601)
  After 500mL; Session 4 | 32.11 (3.216) | 23.11 (4.861)
  After 500mL; Session 5 | 34.67 (5.018) | 21.41 (3.501)
  After 500mL; Session 6 | 32.72 (8.456) | 23.72 (2.967)
  End of session; Session 1 | 26.24 (16.510) | 32.24 (17.922)
  End of session; Session 2 | 27.87 (16.587) | 28.44 (8.748)
  End of session; Session 3 | 19.17 (15.946) | 26.44 (9.281)
  End of session; Session 4 | 28.00 (15.326) | 23.29 (7.928)
  End of session; Session 5 | 30.28 (12.750) | 21.50 (10.671)
  End of session; Session 6 | 28.59 (15.133) | 29.06 (5.043)

ADVERSE EVENTS:
Arm/Group | Secura | Futura
Serious Adverse Events (participants affected / at risk) | 4/18 | 1/18
Other Adverse Events (participants affected / at risk) | 15/18 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Secura (N=18) | Futura (N=18)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0
Bacteremia (Blood and lymphatic system disorders) | 1 (1) | 0
Hyperkalemia (Endocrine disorders) | 1 (1) | 0
Atrial Flutter (Cardiac disorders) | 1 (1) | 0
Myocardial Ischemia (Cardiac disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Secura (N=18) | Futura (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 1 (1) | 0 (0)
malaise (General disorders) | 1 (1) | 0 (0)
bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
bronchitis (Infections and infestations) | 0 (0) | 1 (1)
sinusitis (Infections and infestations) | 1 (1) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
device breakage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
device failure (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
device malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
device occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
breath sounds abnormal (Investigations) | 1 (1) | 0 (0)
serum ferritin decreased (Investigations) | 0 (0) | 1 (1)
hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 1 (1)
sciatica (Nervous system disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Site may publish its own results of the FUTURA Trial after a cooperative publication or 12 months after Sponsor's final evaluation of all the FUTURA Trial data from all sites, whichever occurs first. At least 90 days prior to submitting a manuscript to a publisher or other outside persons or prior to any public presentation, a copy of the abstract, manuscript, or presentation will be provided to Sponsor for review and comment. Sponsor shall have said 90 day period to respond w/ comment.